CLINICAL TRIAL: NCT03848962
Title: iSpecimen Network Protocol: Collection and Distribution of Remnant and Research Use Only Biospecimens for Novel Research Uses
Brief Title: Collection and Distribution of Biospecimens for Novel Research Uses
Status: Recruiting | Type: Observational
Sponsor: iSpecimen Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ISPC-160630-REM/RUO
Record Dates: First submitted 2019-02-11; First posted 2019-02-21 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Cancer; Healthy; Gastrointestinal Complication; Autoimmune Diseases; Infectious Disease; Women's Health: High-Risk Pregnancy; Dermatologic Disease; Blood Disease
MeSH Terms: conditions — Neoplasms; Autoimmune Diseases; Communicable Diseases; Skin Diseases; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects for observational study: Various conditions & healthy subjects

SUMMARY:
iSpecimen aims to create a clinical partner network of hospitals, laboratories, academic institutions, and other healthcare organizations ("institutions") capable of providing researchers and educators ("researchers") with annotated biospecimens for use in biomarker discovery and validation; diagnostic test and instrumentation development and validation; therapeutics development; other medical research including the impact that various specimen collection and handling methods and conditions have on research results; and in education such as researcher or physician training (collectively "research").

DETAILED DESCRIPTION:
The level of involvement for each network institution will vary based on the type of specimen to which they have access (e.g. biofluids, tissues and/or cells) and the category of collection (remnant specimens that were originally collected for clinical testing and/or specimens specifically collected for research) in accordance with the institution's elected preferences.

In most cases, potential participants will be identified and approached upon presenting for clinical care or recruited specifically for the study using outreach programs. If additional screening activities are required to determine eligibility criteria, the potential participant may be presented with the opportunity to participate in these activities as part of the study. These screening activities will be minimal risk in nature and are described further below. Should potential participants meet screening criteria, they may then be asked to provide biospecimens according to current research needs. Individual participants or groups of participants may be sought according to specific clinical, lifestyle, and/or demographic characteristics. The providers of these samples may be healthy participants or participants with a medical condition of interest to the research community but regardless, all specimens collected under this protocol (whether for screening purposes and for distribution to researchers) will qualify as minimal risk activities.

Biospecimens may be distributed to researchers at academic institutions, hospitals, clinical and government laboratories, and corporations including diagnostic, medical device, biopharmaceutical and biotechnology companies. The types of research studies and testing that may be performed using the biospecimens will be varied, and it is not possible to provide a description of all potential studies. Some researchers may perform genetic testing on the specimens, some may use the specimens to develop cell lines, and some may cryopreserve the specimens for many years, awaiting a research use. The specimens may also be used for educational purposes, such as training lab techs on the proper testing of samples or physicians on the proper reading of stained slides. The iSpecimen consent forms will indicate a broad scope of possible research and educational uses and activities.

ELIGIBILITY:
Inclusion Criteria:

* Individual is developmentally aged 7 years old and above for RUO collections (only)
* Individual meets requirements of a current request for research materials from iSpecimen
* If a blood collection will be performed as part of the screening process or RUO collection, the individual's health will be assessed by medical staff through medical record review, clinical exam, and/or the review of an updated medical history as provided by the participant
* Individual has reviewed and signed a consent form for an RUO specimen collection if required as part of the research or if a minor or a person with diminished decision-making capacity, their parent/guardian or Legally Authorized Representative has reviewed and signed the consent form on their behalf.
* Individual has reviewed and signed a consent form for remnant specimen usage in research if required as part of the research or if a minor or a person with diminished decision-making capacity, their parent/guardian or Legally Authorized Representative has reviewed and signed the consent form on their behalf

Exclusion Criteria:

* Subjects that do not meet the inclusion criteria outlined above.

Ages: 1 Month to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: iSpecimen will specify the population for screening and biospecimen collection, based on current research requests submitted to iSpecimen by researchers. All potential participants whose diagnoses, demographic profile, and/or clinically indicated care are consistent with the specified criteria for the collection will be considered eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-06-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Collection of Biospecimens for Novel Research Uses | 10 years
  Repository of diseased and healthy tissue, blood derivatives and related biological specimens

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - iSpecimen, Huntsville, Alabama
  - iSpecimen, Lexington, Massachusetts